CLINICAL TRIAL: NCT01318941
Title: LUMINOUS: Study to Observe the Effectiveness and Safety of Ranibizumab Through Individualized Patient Treatment and Associated Outcomes
Brief Title: Observe the Effectiveness and Safety of Ranibizumab in Real Life Setting
Acronym: LUMINOUS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002A2406
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Wet Age Related Macular Degeneration, Diabetic Macular Edema, Retinal Vein Occlusion; Wet Age Related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
Keywords: Ophthalmology, age-related macular degeneration, Diabetic Macular Edema, Retinal Vein Occlusion, ranibizumab; Ophthalmology; Age-related macular degeneration; Diabetic Macular Edema; Retinal Vein Occlusion; LUMINOUS; Ranibizumab
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ranibizumab
  Interventions: Drug: Ranibizumab; Other: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab
Other: Ranibizumab

SUMMARY:
This study will describe the long-term safety and effectiveness, treatment patterns,and patient reported quality of life associated with ranibizumab treatment in routine clinical practice for all approved indication included in the local product label.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, within age limits as defined by local regulations and local product label, who have previously been treated with, who are currently being treated with or initiating treatment with ranibizumab for any approved indication included in the local product label
* Willing and able to provide informed written consent personally or by legal proxy

Exclusion Criteria:

* Simultaneous participation in a study that includes administration of any investigational drug or procedure
* Systemic or ocular treatment with any VEGF inhibitor other than ranibizumab in the 90 days prior to enrollment
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient ophthalmology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 30490 (Actual)
Dates: Start 2011-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mean Visual Acuity (VA) and mean change in VA | 3,6, and 12 months from the baseline visit, and annually thereafter
Incidence rate, relationship and severity of treatment emergent ocular and non-ocular adverse events | Defined time periods during study duration from FPFV until 30 days after LPLV
Mean visual acuity at quarterly intervals for the primary treated eye set | Quarterly intervals from baseline visit during study duration (5 years)

SECONDARY OUTCOMES:
Incidence rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the time the patient signed the informed consent until 30 days after study discontinuation
Number of ranibizumab injections administered per patient, per eye, and per person-year | annually
"National Eye Institute Visual Functioning Questionnaire-25" change from baseline | annually
Overall number of ranibizumab injections, number of visits, time interval between injections, duration of treatment, number of re-treatment, and reasons for treatment termination | Over time during study duration (5 years)
Change from baseline in National Eye Institute Visual Function Questionnaire 25 composite and sub-scale scores | Over time during study duration (5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (409):
- Argentina (15):
  - Novartis Investigative Site, Buenos Aires, Argentina
  - Novartis Investigative Site, Concepción del Uruguay, Argentina
  - Novartis Investigative Site, Córdoba, Argentina
  - Novartis Investigative Site, Guaymallén, Mendoza, Argentina
  - Novartis Investigative Site, Rosario, Argentina
  - Novartis Investigative Site, San Martin, Buenos Aires, Argentina
  - Novartis Investigative Site, Santa Fe, Argentina
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Caballito
  - Novartis Investigative Site, Ciudad de Buenos Aires,
  - Novartis Investigative Site, La Plata
  - Novartis Investigative Site, Santa Fe
- Australia (20):
  - Novartis Investigative Site, Chatswood, New South Wales
  - Novartis Investigative Site, Forster, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, North Ryde, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Strathfield, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Brisbane, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, North Adelaide, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, South Launceston, Tasmania
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Glen Waverley, Victoria
  - Novartis Investigative Site, Oakleigh, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (15):
  - Novartis Investigative Site, Aalst, Belgium
  - Novartis Investigative Site, Aarschot, Belgium
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Dinant
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Mouscron
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Nivelles
  - Novartis Investigative Site, Reet
  - Novartis Investigative Site, Yvoir
  - Novartis Investigative Site, Zottegem
- Brazil (6):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (17):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Miramichi, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Downsview, Ontario
  - Novartis Investigative Site, East Brockville, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Vaughan, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Barrie
  - Novartis Investigative Site, Drummondville
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Ontario
- Novartis Investigative Site, Calama, Chile
- China (13):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Guiyang, Guizhou
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Changchun
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Fujian
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Ürümqi
- Colombia (5):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Armenia, Quindío Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Yopal
- Novartis Investigative Site, San José, Costa Rica, Costa Rica
- Czechia (7):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava-Poruba
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Ustri Nad Labem
- Novartis Investigative Site, Santo Domingo, Republica Dominicana, Dominican Republic
- Novartis Investigative Site, Ciudadela Kennedy, Guayaquil, Ecuador
- Egypt (2):
  - Novartis Investigative Site, Cairo, Cairo Governorate
  - Novartis Investigative Site, Giza
- France (14):
  - Novartis Investigative Site, Poitiers, France
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Melun
  - Novartis Investigative Site, Montargis
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vannes
- Germany (16):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dannenberg
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ingolstadt
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rothenburg
  - Novartis Investigative Site, Schriesheim
  - Novartis Investigative Site, Tönisvorst
  - Novartis Investigative Site, Tübingen
- Greece (10):
  - Novartis Investigative Site, Alexandroupoli, Greece
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion - Crete, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Patra - RIO, GR
  - Novartis Investigative Site, Rethymno, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Lamia, Phthiotis
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Novartis Investigative Site, Kowloon, Hong Kong, Hong Kong
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- India (6):
  - Novartis Investigative Site, Pātia, Bhudaneswar
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, New Delhi
- Ireland (2):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Waterford
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (9):
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Alessandria
  - Novartis Investigative Site, Belluno
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Reggio Calabria
  - Novartis Investigative Site, Roma
- Japan (83):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Aomori, Aomori
  - Novartis Investigative Site, Sakura, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Yoshida-gun, Fukui
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Inashiki-gun, Ibaraki
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Ashigarakami-gun, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Yokohama, Kangawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyakonojō, Miyazaki
  - Novartis Investigative Site, Miyazaki, Miyazaki
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Izunokuni, Shizuoka
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Shimotsuka-gun, Tochigi
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Urayasu, Tokyo
  - Novartis Investigative Site, Imizu-shi, Toyama
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Chiyoda-ku
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Hamamatsu
  - Novartis Investigative Site, Hokkaido
  - Novartis Investigative Site, Hyōgo
  - Novartis Investigative Site, Ishikawa
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Kakogawa-shi
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Kawasaki-shi
  - Novartis Investigative Site, Kitami-shi
  - Novartis Investigative Site, Koriyama-shi
  - Novartis Investigative Site, Kouchi
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Nagano
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Nantan-shi
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōtsu
  - Novartis Investigative Site, Saitama-ken
  - Novartis Investigative Site, Sanjo-shi
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Shunan-shi
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Toyohashi
  - Novartis Investigative Site, Wakayama
  - Novartis Investigative Site, Yamagata
- Malaysia (2):
  - Novartis Investigative Site, Batu Caves, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (5):
  - Novartis Investigative Site, Col. Lomas de Chapultepec, CP
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterray, Nuevo León
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mérida, Yucatán
- Netherlands (3):
  - Novartis Investigative Site, Almere Stad
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Tilburg
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Peru (3):
  - Novartis Investigative Site, Lima, Lima Province
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
- Poland (14):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Chojnice
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gda¿sk
  - Novartis Investigative Site, Kalisz
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wałbrzych
  - Novartis Investigative Site, Wołomin
- Portugal (6):
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Aveiro
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Santa Maria da Feira
- Russia (18):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Chita
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Khabarovsk
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Surgut
  - Novartis Investigative Site, Tambov
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yakutsk
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- Slovakia (11):
  - Novartis Investigative Site, Banksa Bystrica, Slovak Republic
  - Novartis Investigative Site, Trebišov, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Nové Zámky, Slovakia
  - Novartis Investigative Site, Zvolen, Slovakia
  - Novartis Investigative Site, Žilina, Slovakia
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Ružomberok
  - Novartis Investigative Site, Trenčín
- Slovenia (4):
  - Novartis Investigative Site, Novo Mesto, Slovenia
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Maribor
- South Korea (8):
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (17):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Logroño, Hospital La Rioja Provincia
  - Novartis Investigative Site, Murcia, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Zaragoza, Zaragoza
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Granollers
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Altindag / Ankara
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Mecidiyekoy/Istanbul
- Ukraine (4):
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Luhansk
  - Novartis Investigative Site, Odesa
- United Kingdom (46):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Durham, County Durham
  - Novartis Investigative Site, Torquay, Devon,
  - Novartis Investigative Site, Bolton, England
  - Novartis Investigative Site, Solihull, England
  - Novartis Investigative Site, Southampton, England
  - Novartis Investigative Site, Wakefield, England
  - Novartis Investigative Site, Belfast, Essex
  - Novartis Investigative Site, Romford, Essex
  - Novartis Investigative Site, Cheltenham, Gloucestershire
  - Novartis Investigative Site, Blackburn, Lancashire
  - Novartis Investigative Site, Hull, Lancashire
  - Novartis Investigative Site, Leicester, Lancashire
  - Novartis Investigative Site, Coventry, London
  - Novartis Investigative Site, Derby, London
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Oxford, Oxfordshire
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Worcester, UK
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Bedford
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Inverness
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Maidstone
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Merseyside
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Southend
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Uxbridge
  - Novartis Investigative Site, Wolverhampton
  - Novartis Investigative Site, York
- Venezuela (5):
  - Novartis Investigative Site, Porlamar Local 02, Isla Margarita
  - Novartis Investigative Site, Caracas
  - Novartis Investigative Site, Caracas, Piso 6, Ofic. 607
  - Novartis Investigative Site, Santa Paula
  - Novartis Investigative Site, Torre Venezuela, Piso 1

REFERENCES:
- [Derived] Holz FG, Minnella AM, Tuli R, Yoganathan P, Parikh S, Hamilton R; LUMINOUS study group. Ranibizumab treatment patterns in prior ranibizumab-treated neovascular age-related macular degeneration patients: Real-world outcomes from the LUMINOUS study. PLoS One. 2020 Dec 30;15(12):e0244183. doi: 10.1371/journal.pone.0244183. eCollection 2020. PMID 33378369
- [Derived] Leys AM, Ramboer E, Favreau M, Denhaerynck K, MacDonald K, Abraham I, Brie H. Long-Term Ranibizumab Treatment in Neovascular Age-Related Macular Degeneration: A Belgian Subanalysis from the Global Real-World LUMINOUSTM Study. Clin Ophthalmol. 2020 Jun 2;14:1473-1481. doi: 10.2147/OPTH.S242547. eCollection 2020. PMID 32581505
- [Derived] Pearce I, Clemens A, Brent MH, Lu L, Gallego-Pinazo R, Minnella AM, Creuzot-Garcher C, Spital G, Sakamoto T, Dunger-Baldauf C, McAllister IL; all the LUMINOUS study investigators. Real-world outcomes with ranibizumab in branch retinal vein occlusion: The prospective, global, LUMINOUS study. PLoS One. 2020 Jun 18;15(6):e0234739. doi: 10.1371/journal.pone.0234739. eCollection 2020. PMID 32555630
- [Derived] Mitchell P, Sheidow TG, Farah ME, Mahmood S, Minnella AM, Eter N, Eldem B, Al-Dhibi H, Macfadden W, Parikh S, Dunger-Baldauf C, Mahgoub MM, Schmidt-Erfurth U; LUMINOUS study investigators. Effectiveness and safety of ranibizumab 0.5 mg in treatment-naive patients with diabetic macular edema: Results from the real-world global LUMINOUS study. PLoS One. 2020 Jun 3;15(6):e0233595. doi: 10.1371/journal.pone.0233595. eCollection 2020. PMID 32492069
- [Derived] Schmidt-Erfurth U, Chong V, Loewenstein A, Larsen M, Souied E, Schlingemann R, Eldem B, Mones J, Richard G, Bandello F; European Society of Retina Specialists. Guidelines for the management of neovascular age-related macular degeneration by the European Society of Retina Specialists (EURETINA). Br J Ophthalmol. 2014 Sep;98(9):1144-67. doi: 10.1136/bjophthalmol-2014-305702. PMID 25136079